CLINICAL TRIAL: NCT06179264
Title: Preliminary Evaluation of an Online Acceptance and Commitment Training Program for Individuals with Chronic Health Conditions
Brief Title: Evaluating an Online Acceptance and Commitment Training Program for Individuals with Chronic Health Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Professor of Psychology, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB: #13890
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Stress, Psychological; Depression; Well-Being, Psychological
Keywords: acceptance and commitment therapy; chronic health conditions
MeSH Terms: conditions — Stress, Psychological; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized wait list control trial. Parallel assignment of participants to treatment and wait list groups. Wait list participants receive treatment after 10 weeks of waiting. Treatment participants receive treatment immediately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Following random assignment to the condition after completing baseline assessment, participants will be instructed to complete the ACT Guide for Chronic Health Conditions program over the next 6 weeks.
  Interventions: Behavioral: ACT Guide for Chronic Health Conditions
- Waitlist Control (No Intervention): Following random assignment to the condition after completing baseline assessment, participants will be instructed to wait to receive the intervention after a period of 10 weeks (this accounts for the 6 weeks that treatment condition participants are given to complete the program, plus the 4 interim between post-assessment and follow-up.

INTERVENTIONS:
Behavioral: ACT Guide for Chronic Health Conditions — Acceptance and commitment therapy (ACT) combines the skills of acceptance, cognitive defusion, being present, self as context, values, and committed action to help individuals engage with a meaningful life. The current project is an online, self-guided, 6-session intervention based on ACT. The program is intended to help individuals with chronic health conditions improve their quality of life and mental health. Each session is expected to take about 30 minutes each, and the entire program will take 6 weeks to complete, as users will be encouraged to work on one session per week. Within each session, participants will read about concepts and ACT metaphors, apply ACT concepts to general and chronic health condition specific vignettes, and apply ACT concepts to their own lives and situations related to their chronic health condition. Interactive experiences are included in each session and ends with a printable summary with practice skills before proceeding.
  Arms: Treatment

SUMMARY:
Chronic health conditions (CHC) commonly share the challenge of impaired health-related quality of life, negatively impacting the lives of millions of people in the United States. Long term effects for living with a chronic health condition are likely to include poor self-management behaviors, which are related to avoidance of disease related thoughts and feelings (e.g., health anxiety) and can be addressed directly with psychosocial interventions. With the focus on fostering values driven and meaningful behavior while accepting thoughts and feelings, ACT may prove to be a particularly effective approach for individuals coping with the challenging symptoms and effects of having a chronic health condition. Previous web-based ACT interventions for CHCs have focused on building ACT skills for a narrow subset of CHCs (e.g., breast cancer, diabetes, tinnitus). While there is added benefit for a self-help program for populations with specific stressors or conditions, there is also a high prevalence of comorbidity in CHCs, shared challenges in illness management and coping, and clear evidence that ACT works effectively across CHCs to improve quality of life. Thus, our goal of this research project is to evaluate a new 6 session, online, self-guided ACT program for adults with chronic health conditions broadly to improve their quality of life and wellbeing through a randomized controlled trial. The specific aims are:

1. To evaluate the feasibility of an initial prototype of ACT program for adults with CHC's as indicated by recruitment, retention, and adherence rates.
2. To evaluate the acceptability as indicated by self-reported program satisfaction and qualitative feedback following the course completion.
3. To identify ways to further refine the program based on participant self-reported satisfaction with sessions and open-ended text-based feedback.
4. To test the efficacy of the program on improving quality of life among adults with CHC's.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Currently living in the U.S.
* Self-report having at least 1 chronic health condition (e.g., cardiovascular disease, cancer, diabetes, chronic pain, rheumatoid arthritis, HIV, Parkinson's disease, irritable bowel syndrome, Crohn's disease, chronic obstructive pulmonary disease, multiple sclerosis)
* Self-report having had the chronic health condition for ≥ 3 months
* Can access the internet via computer, mobile phone, or tablet
* Have an interest in using an online mental health intervention

Exclusion Criteria:

• Not fluent in reading English (at this point the online program can only be feasibly and competently delivered in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Mental Health Continuum - Short Form (MHC-SF; to assess positive mental health) | baseline, post-assessment (6 weeks after baseline), follow-up (10 weeks after baseline)
  This 14-item measure assesses positive mental health, with a total score as well as subscales for emotional, psychological and social wellbeing. The scale uses 6-point Likert scale ranging from 0 "never" to 5 "everyday." Items are summed, yielding a total score ranging from 0 to 70. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
CompACT (to assess psychological flexibility) | baseline, post-assessment (6 weeks after baseline), follow-up (10 weeks after baseline)
  This 23-item measure will be used to measure the ACT process of change, psychological flexibility, including subscales for openness to experience, behavioral awareness, and valued action. The CompACT will serve as the primary outcome for this study in order to test whether a single session intervention is sufficient to target the ACT process of change of psychological flexibility. The scale uses 7-point Likert scale ranging from 0 to 6, with total score ranging from 0 to 138. A higher score indicates a better outcome.
Work and Social Adjustment Scale (WSAS; to assess psychosocial functioning as impacted by chronic health conditions) | baseline, post-assessment (6 weeks after baseline), follow-up (10 weeks after baseline)
  The 5-item Work and Social Adjustment Scale (WSAS; Mundt et al., 2002) assesses the degree to which chronic health conditions interfere with psychosocial functioning (e.g., ability to work, complete home tasks). The scale uses 9-point Likert scale ranging from 0 to 8, with total score ranging from 0 to 40. A higher score indicates a worse outcome.
Depression, Anxiety and Stress Scale (DASS-21) | baseline, post-assessment (6 weeks after baseline), follow-up (10 weeks after baseline)
  This 21-item measure will be used to assess the subscales of depression, anxiety, and stress, with a total score representing overall psychological distress. The scale uses 4-point Likert scale ranging from 0 to 3. To calculate the total score, the score for each individual item is doubled. The total score ranges from 0 to 126, and each of the three subscales ranges from 0 to 42. A higher score indicates a worse outcome.
Program satisfaction (Responses to a series of single item Likert-scale items about satisfaction with the intervention) | post-assessment (6 weeks after baseline)
  A series of program satisfaction items will be asked in the ACT condition immediately post-intervention and at 1-week and 1-month follow up based on items used in our previous online ACT trials. This will include a series of items assessing features of program satisfaction (e.g., overall satisfaction, helpfulness, perceived fit, if the program was too short or long, etc…) on a scale from 1 (strongly disagree) to 6 (strongly agree). These are not intended to be summed for a total score. Whether a higher or lower score is more desirable depends on the individual item.
  In addition, participants will be asked to type responses to open ended questions assessing what they learned from the program and areas needing further revision.
System usability scale (SUS; to measure program usability) | post-assessment (6 weeks after baseline)
  At posttreatment only, participants will be asked to rate their perception of the ACT program's usability using the System Usability Scale. This measure consists of 10 items assessing program usability. The scale uses 5-point Likert scale ranging from 1 to 5. Scores are transformed to be on a scale that ranges from 0 to 100. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Levin, PhD, Principal Investigator — Utah State University; Ty B Aller, Study Director — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Dr. Michael Levin or Dr. Aller will review requests and criteria.

REFERENCES:
- [Background] Dindo L, Van Liew JR, Arch JJ. Acceptance and Commitment Therapy: A Transdiagnostic Behavioral Intervention for Mental Health and Medical Conditions. Neurotherapeutics. 2017 Jul;14(3):546-553. doi: 10.1007/s13311-017-0521-3. PMID 28271287
- [Background] Feliu-Soler A, Montesinos F, Gutierrez-Martinez O, Scott W, McCracken LM, Luciano JV. Current status of acceptance and commitment therapy for chronic pain: a narrative review. J Pain Res. 2018 Oct 2;11:2145-2159. doi: 10.2147/JPR.S144631. eCollection 2018. PMID 30323649
- [Background] Grady PA, Gough LL. Self-management: a comprehensive approach to management of chronic conditions. Am J Public Health. 2014 Aug;104(8):e25-31. doi: 10.2105/AJPH.2014.302041. Epub 2014 Jun 12. PMID 24922170
- [Background] Graham CD, Gouick J, Krahe C, Gillanders D. A systematic review of the use of Acceptance and Commitment Therapy (ACT) in chronic disease and long-term conditions. Clin Psychol Rev. 2016 Jun;46:46-58. doi: 10.1016/j.cpr.2016.04.009. Epub 2016 Apr 20. PMID 27176925
- [Background] Herbert MS, Dochat C, Wooldridge JS, Materna K, Blanco BH, Tynan M, Lee MW, Gasperi M, Camodeca A, Harris D, Afari N. Technology-supported Acceptance and Commitment Therapy for chronic health conditions: A systematic review and meta-analysis. Behav Res Ther. 2022 Jan;148:103995. doi: 10.1016/j.brat.2021.103995. Epub 2021 Nov 12. PMID 34800873
- [Background] Samiei Siboni F, Alimoradi Z, Atashi V, Alipour M, Khatooni M. Quality of Life in Different Chronic Diseases and Its Related Factors. Int J Prev Med. 2019 May 17;10:65. doi: 10.4103/ijpvm.IJPVM_429_17. eCollection 2019. PMID 31198500
- [Background] Bangor, A., Kortum, P. T., & Miller, J. T. (2008). An empirical evaluation of the system usability scale. Intl. Journal of Human-Computer Interaction, 24(6), 574-594.
- [Background] Francis, A. W., Dawson, D. L., & Golijani-Moghaddam, N. (2016). The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of Contextual Behavioral Science, 5(3), 134-145.
- [Background] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Derived] Levin ME, Aller TB, Klimczak KS, Donahue ML, Knudsen FM. Digital acceptance and commitment therapy for adults with chronic health conditions: Results from a waitlist-controlled trial. Behav Res Ther. 2025 May;188:104729. doi: 10.1016/j.brat.2025.104729. Epub 2025 Mar 16. PMID 40120228